CLINICAL TRIAL: NCT04892914
Title: Feasibility of the Embr Thermal Device for Management of Hot Flashes in Men With Prostate Cancer
Brief Title: Embr Thermal Device for Hot Flash Management in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Embr Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMBR-PC-001
Record Dates: First submitted 2021-05-11; First posted 2021-05-19 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer; Hot Flashes
Keywords: androgen deprivation therapy; orchiectomy; prostate carcinoma; night sweats; hormone therapy
MeSH Terms: conditions — Prostatic Neoplasms; Hot Flashes

STUDY DESIGN:
Intervention Model Description: Embr thermal device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embr thermal device (Experimental): Use of the Embr thermal device
  Interventions: Device: Embr thermal device

INTERVENTIONS:
Device: Embr thermal device — Participants use the Embr thermal device for 4 weeks

SUMMARY:
This study is being conducted to evaluate if the Embr thermal device is useful for men who experience bothersome hot flashes as a result of prostate cancer treatment.

DETAILED DESCRIPTION:
The Embr thermal device is a smart device that is worn on the inside of the wrist. It is about the size of a smart watch. The Embr thermal device produces cooling or warming temperature sensations that make some people feel slightly cooler or warmer. This objective of this study is to evaluate if the Embr thermal device is useful for men who experience bothersome hot flashes as a result of prostate cancer treatment. The study will take place over 4 weeks. The primary outcome is feasibility of the Embr thermal device in men with prostate cancer. Secondary outcomes include preliminary efficacy of the device, which will include the change in hot flash interference sleep measures (sleep impairment and fatigue). This is a remote study--all study assessments will be completed electronically.

ELIGIBILITY:
Inclusion Criteria:

* Have received a diagnosis of prostate cancer and have received treatment with GnRH agonist or antagonist therapy or orchiectomy at least 1 month prior to enrollment.
* May have received prior definitive radiation therapy or surgery (>60 days prior to study).
* Have bothersome hot flashes (occurrence ≥ 28 times per week and at least moderately bothersome).
* Presence of hot flashes for >30 days prior to study entry.
* Have a working smartphone (iPhone 6 or greater; or Android 8.0 or greater).
* Willing to downloading and use the Embr thermal device companion app on their phone
* Willing to wear the Embr thermal device for 4 weeks, and charge and sync the device daily
* In order to complete the mandatory patient-completed measures, participants must be able to speak and/or read English

Exclusion Criteria:

* Planned treatment with chemotherapy and/or any medical intervention that will impact hot flashes, sleep, or other daily activities of daily life during the 4-week study.
* History of a known sleep disorder, other than insomnia (eg, obstructive sleep apnea, restless leg syndrome), or medical or psychiatric condition that affects sleep, or undergoing treatment for insomnia.
* History of cognitive impairment or dysfunction.
* Seizure history, history of recurrent falls, or known brain metastases.
* Uncontrolled intercurrent illness.
* Individuals with a second malignancy other than non-melanoma skin cancers.
* Individuals taking psychotropic medications or illicit drugs that may alter cognition, concentration, or behavior.
* Individuals taking prescription sleep medications.
* Individuals who report consuming more than 7 alcoholic beverages/week and/or frequent alcohol consumption within 2 hours prior to bed.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Embr thermal device usage, average number of minutes per day per participant | Weeks 0 to 4
  Number of minutes logged with the Embr device.
Embr thermal device usage, average number of sessions per day per participant | Weeks 0 to 4
  Number of sessions logged with the Embr device.

SECONDARY OUTCOMES:
Hot Flash Related Daily Interference Scale (HFRDIS), change in score | Week 0, 2, 4
  The Hot Flash Related Daily Interference Scale is a 10-item self-report measure that assesses the interference on several aspects of functioning associated with hot flashes. This valid and reliable self-report measure is widely used in prostate cancer research. Scores range from 0 to 100, with higher scores indicating greater interference.
PROMIS Sleep Disturbance short form 4a, change in score | Week 0, 2, 4
  The PROMIS Sleep Disturbance SF 4a is a 4-item self report measure of perceived difficulties falling asleep and staying asleep, as well as sleep satisfaction. The 4 items are scored 1-5 where 1 is good quality and 5 is poor quality for a total score range of 4 (good quality) to 20 (poor quality).
PROMIS Sleep-Related Impairment short form 8a, change in score | Weeks 0, 2, 4
  The PROMIS Sleep-Related Impairment SF 8a is an 8-item self reported measure of perceived alertness, sleepiness, and tiredness during usual waking hours. The 8 items are scored 1-5 where 1 is good quality and 5 is poor quality for a total score range of 8 (good quality) to 40 (poor quality).
Epworth sleepiness scale, change in score | Week 0, 2, 4
  The Epworth Sleepiness Scale is a widely used measure of daytime sleepiness. Scores range from 0 to 24; scores of greater than 10 indicate excessive daytime sleepiness.

OTHER OUTCOMES:
Vasomotor Symptom Survey | Week 0, 1, 2, 3, 4
  Self-report 10-question survey of hot flash and night sweat number, duration, interference, bothersome rating, and control of interference. Score range 0 to 86 with higher score indicating greater negative impact of vasomotor symptoms.
Temperature-related quality of life and symptoms, change in score | Week 0, 2, 4
  Self-report measure of temperature-related quality of life and symptoms. Scores range from 0 to 100 with higher scores indicating greater quality of life.
User acceptance | Week 4
  Self-report 8-question survey at end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Morgans, MD, MPH, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Embr Labs (Remote study site), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized dataset of selected variables that underlie results in a publication. Some data may not be amenable to complete anonymization and will not be shared to ensure appropriate confidentiality of participant's data.
Time Frame: Beginning 6 months after publication
Access Criteria: Upon appropriate data request